CLINICAL TRIAL: NCT00556270
Title: Matrifen for Therapy of Severe, Chronic Pain.
Brief Title: Efficacy of Matrifen in Patients Older Than 18 Years With Severe, Chronic Pain
Acronym: MATRIX II
Status: Completed | Type: Observational
Sponsor: Nycomed (Industry)
Other Study IDs: Matri Matrix II 07/10
Record Dates: First submitted 2007-11-08; First posted 2007-11-09 (Estimated); Last update posted 2012-05-07 (Estimated); Status verified 2012-05

CONDITIONS: Severe, Chronic Pain
Keywords: pain; fentanyl; transdermal patch
MeSH Terms: conditions — Chronic Pain; Pain | interventions — Fentanyl

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Matrix II
  Interventions: Drug: Matrifen

INTERVENTIONS:
Drug: Matrifen — as defined in the Summary of Product Characteristics (Fachinformation Chapter 4.2)

SUMMARY:
The aim of the study is to evaluate the efficacy and safety of matrifen in patients with severe and chronic pain who can only be sufficiently treated with opioid analgesics (WHO class 3).

ELIGIBILITY:
Main inclusion criteria:

* Patients with severe, chronic pain

Main exclusion criteria:

* Hypersensitivity of fentanyl
* Co-administration of monoaminooxidase-inhibitors
* Pregnancy
* Respiratory depression
* Chronic obstructive pulmonary disease (COPD)
* Drug abuse
* Impairment of CNS functions
* Other criteria as defined in the Summary of Product Characteristics (Fachinformation Chapter 4.3)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Outpatients
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2007-11; Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Treatment success, efficacy of Matrifen | within 1 month

SECONDARY OUTCOMES:
Safety and tolerability of fentanyl and the transdermal system, quality of life | within 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Thomas D. Bethke, PhD, MD, Study Director — Nycomed Deutschland GmbH, 78467 Konstanz, Germany
Locations (617):
- Germany (617):
  - "Nycomed Deutschland GmbH", Aachen
  - "Nycomed Deutschland GmbH", Aalen
  - "Nycomed Deutschland GmbH", Achim
  - "Nycomed Deutschland GmbH", Ahaus
  - "Nycomed Deutschland GmbH", Ahlen
  - "Nycomed Deutschland GmbH", Aicha
  - "Nycomed Deutschland GmbH", Albstadt
  - "Nycomed Deutschland GmbH", Alfeld
  - "Nycomed Deutschland GmbH", Alfhausen
  - "Nycomed Deutschland GmbH", Altdorf
  - "Nycomed Deutschland GmbH", Altenburg
  - "Nycomed Deutschland GmbH", Altenstadt
  - "Nycomed Deutschland GmbH", Altlußheim
  - "Nycomed Deutschland GmbH", Alzenau in Unterfranken
  - "Nycomed Deutschland GmbH", Amorbach
  - "Nycomed Deutschland GmbH", Angermünde
  - "Nycomed Deutschland GmbH", Anklam
  - "Nycomed Deutschland GmbH", Annweiler am Trifels
  - "Nycomed Deutschland GmbH", Ansbach
  - "Nycomed Deutschland GmbH", Apolda
  - "Nycomed Deutschland GmbH", Arnsberg
  - "Nycomed Deutschland GmbH", Arnsdorf
  - "Nycomed Deutschland GmbH", Arnstadt
  - "Nycomed Deutschland GmbH", Aschendorf
  - "Nycomed Deutschland GmbH", Attenkirchen
  - "Nycomed Deutschland GmbH", Aue
  - "Nycomed Deutschland GmbH", Auerbach
  - "Nycomed Deutschland GmbH", Augsburg
  - "Nycomed Deutschland GmbH", Aumühle
  - "Nycomed Deutschland GmbH", Aurich
  - "Nycomed Deutschland GmbH", Aßlar
  - "Nycomed Deutschland GmbH", Bad Arolsen
  - "Nycomed Deutschland GmbH", Bad Bederkesa
  - "Nycomed Deutschland GmbH", Bad Berka
  - "Nycomed Deutschland GmbH", Bad Bevensen
  - "Nycomed Deutschland GmbH", Bad Dürrenberg
  - "Nycomed Deutschland GmbH", Bad Dürrheim
  - "Nycomed Deutschland GmbH", Bad Ems
  - "Nycomed Deutschland GmbH", Bad Essen
  - "Nycomed Deutschland GmbH", Bad Fallingbostel
  - "Nycomed Deutschland GmbH", Bad Frankenhausen
  - "Nycomed Deutschland GmbH", Bad Hersfeld
  - "Nycomed Deutschland GmbH", Bad Krozingen
  - "Nycomed Deutschland GmbH", Bad Langensalza
  - "Nycomed Deutschland GmbH", Bad Lauterberg im Harz
  - "Nycomed Deutschland GmbH", Bad Liebenwerda
  - "Nycomed Deutschland GmbH", Bad Lippspringe
  - "Nycomed Deutschland GmbH", Bad Marienberg
  - "Nycomed Deutschland GmbH", Bad Oeynhausen
  - "Nycomed Deutschland GmbH", Bad Oldesloe
  - "Nycomed Deutschland GmbH", Bad Pyrmont
  - "Nycomed Deutschland GmbH", Bad Sachsa
  - "Nycomed Deutschland GmbH", Bad Salzuflen
  - "Nycomed Deutschland GmbH", Bad Salzungen
  - "Nycomed Deutschland GmbH", Bad Schwalbach
  - "Nycomed Deutschland GmbH", Bad Tennstedt
  - "Nycomed Deutschland GmbH", Bahrdorf
  - "Nycomed Deutschland GmbH", Balingen
  - "Nycomed Deutschland GmbH", Ballstädt
  - "Nycomed Deutschland GmbH", Bamberg
  - "Nycomed Deutschland GmbH", Bargstedt
  - "Nycomed Deutschland GmbH", Barnstädt
  - "Nycomed Deutschland GmbH", Barsinghausen
  - "Nycomed Deutschland GmbH", Bergfelde
  - "Nycomed Deutschland GmbH", Bergisch Gladbach
  - "Nycomed Deutschland GmbH", Bergrheinfeld
  - "Nycomed Deutschland GmbH", Berlin
  - "Nycomed Deutschland GmbH", Berne
  - "Nycomed Deutschland GmbH", Bevern
  - "Nycomed Deutschland GmbH", Beverungen
  - "Nycomed Deutschland GmbH", Biberach
  - "Nycomed Deutschland GmbH", Bielefeld
  - "Nycomed Deutschland GmbH", Bischofswerda
  - "Nycomed Deutschland GmbH", Bisingen
  - "Nycomed Deutschland GmbH", Bitburg
  - "Nycomed Deutschland GmbH", Blankenburg
  - "Nycomed Deutschland GmbH", Bobenheim-Roxheim
  - "Nycomed Deutschland GmbH", Bobritzsch
  - "Nycomed Deutschland GmbH", Bochum
  - "Nycomed Deutschland GmbH", Bockau
  - "Nycomed Deutschland GmbH", Bohmte
  - "Nycomed Deutschland GmbH", Bottrop
  - "Nycomed Deutschland GmbH", Böhlen
  - "Nycomed Deutschland GmbH", Bramsche
  - "Nycomed Deutschland GmbH", Brand-Erbisdorf
  - "Nycomed Deutschland GmbH", Braunsbedra
  - "Nycomed Deutschland GmbH", Braunschweig
  - "Nycomed Deutschland GmbH", Bredstedt
  - "Nycomed Deutschland GmbH", Breidenbach
  - "Nycomed Deutschland GmbH", Breitenfelde
  - "Nycomed Deutschland GmbH", Bremen
  - "Nycomed Deutschland GmbH", Bremerhaven
  - "Nycomed Deutschland GmbH", Brüel
  - "Nycomed Deutschland GmbH", Burg
  - "Nycomed Deutschland GmbH", Burgdorf, Hanover
  - "Nycomed Deutschland GmbH", Burgstädt
  - "Nycomed Deutschland GmbH", Burkhardtsdorf
  - "Nycomed Deutschland GmbH", Burscheid
  - "Nycomed Deutschland GmbH", Bückeburg
  - "Nycomed Deutschland GmbH", Bünde
  - "Nycomed Deutschland GmbH", Castrop-Rauxel
  - "Nycomed Deutschland GmbH", Celle
  - "Nycomed Deutschland GmbH", Chemnitz
  - "Nycomed Deutschland GmbH", Coesfeld
  - "Nycomed Deutschland GmbH", Cologne
  - "Nycomed Deutschland GmbH", Coswig
  - "Nycomed Deutschland GmbH", Cottbus
  - "Nycomed Deutschland GmbH", Cuxhaven
  - "Nycomed Deutschland GmbH", Dabel
  - "Nycomed Deutschland GmbH", Darmstadt
  - "Nycomed Deutschland GmbH", Daun
  - "Nycomed Deutschland GmbH", Dautphetal
  - "Nycomed Deutschland GmbH", Delitzsch
  - "Nycomed Deutschland GmbH", Demmin
  - "Nycomed Deutschland GmbH", Denkendorf
  - "Nycomed Deutschland GmbH", Denzlingen
  - "Nycomed Deutschland GmbH", Dessau
  - "Nycomed Deutschland GmbH", Dettenheim
  - "Nycomed Deutschland GmbH", Diepholz
  - "Nycomed Deutschland GmbH", Dingolfing
  - "Nycomed Deutschland GmbH", Dorsten
  - "Nycomed Deutschland GmbH", Dortmund
  - "Nycomed Deutschland GmbH", Dörentrup
  - "Nycomed Deutschland GmbH", Dörzbach
  - "Nycomed Deutschland GmbH", Dresden
  - "Nycomed Deutschland GmbH", Ducherow
  - "Nycomed Deutschland GmbH", Dudenhofen
  - "Nycomed Deutschland GmbH", Duisburg
  - "Nycomed Deutschland GmbH", Durmersheim
  - "Nycomed Deutschland GmbH", Dürrröhrsdorf
  - "Nycomed Deutschland GmbH", Düsseldorf
  - "Nycomed Deutschland GmbH", Ebeleben
  - "Nycomed Deutschland GmbH", Eberbach
  - "Nycomed Deutschland GmbH", Ebersbach
  - "Nycomed Deutschland GmbH", Eberstadt
  - "Nycomed Deutschland GmbH", Eberswalde
  - "Nycomed Deutschland GmbH", Eddelak
  - "Nycomed Deutschland GmbH", Edenkoben
  - "Nycomed Deutschland GmbH", Ehra-Lessien
  - "Nycomed Deutschland GmbH", Eimsheim
  - "Nycomed Deutschland GmbH", Eisenach
  - "Nycomed Deutschland GmbH", Eisenberg
  - "Nycomed Deutschland GmbH", Eisenhüttenstadt
  - "Nycomed Deutschland GmbH", Eisleben Lutherstadt
  - "Nycomed Deutschland GmbH", Eiterfeld
  - "Nycomed Deutschland GmbH", Ellefeld
  - "Nycomed Deutschland GmbH", Ellerstadt
  - "Nycomed Deutschland GmbH", Ellwangen
  - "Nycomed Deutschland GmbH", Elstra
  - "Nycomed Deutschland GmbH", Elterlein
  - "Nycomed Deutschland GmbH", Emleben
  - "Nycomed Deutschland GmbH", Emsdetten
  - "Nycomed Deutschland GmbH", Emstek
  - "Nycomed Deutschland GmbH", Engelskirchen
  - "Nycomed Deutschland GmbH", Enger
  - "Nycomed Deutschland GmbH", Eningen unter Achalm
  - "Nycomed Deutschland GmbH", Enkirch
  - "Nycomed Deutschland GmbH", Ennepetal
  - "Nycomed Deutschland GmbH", Eppstein
  - "Nycomed Deutschland GmbH", Erfurt
  - "Nycomed Deutschland GmbH", Eschelbronn
  - "Nycomed Deutschland GmbH", Eschwege
  - "Nycomed Deutschland GmbH", Esens
  - "Nycomed Deutschland GmbH", Espelkamp
  - "Nycomed Deutschland GmbH", Essen
  - "Nycomed Deutschland GmbH", Falkensee
  - "Nycomed Deutschland GmbH", Fehrbellin
  - "Nycomed Deutschland GmbH", Finsterwalde
  - "Nycomed Deutschland GmbH", Floh-Seligenthal
  - "Nycomed Deutschland GmbH", Flonheim
  - "Nycomed Deutschland GmbH", Framersheim
  - "Nycomed Deutschland GmbH", Frankenberg
  - "Nycomed Deutschland GmbH", Frankfurt
  - "Nycomed Deutschland GmbH", Freiberg
  - "Nycomed Deutschland GmbH", Freiburg im Breisgau
  - "Nycomed Deutschland GmbH", Freising
  - "Nycomed Deutschland GmbH", Freyburg
  - "Nycomed Deutschland GmbH", Friedeburg
  - "Nycomed Deutschland GmbH", Friedrichshafen
  - "Nycomed Deutschland GmbH", Friedrichsthal
  - "Nycomed Deutschland GmbH", Furth im Wald
  - "Nycomed Deutschland GmbH", Fürstenberg
  - "Nycomed Deutschland GmbH", Fürstenwalde
  - "Nycomed Deutschland GmbH", Garbsen
  - "Nycomed Deutschland GmbH", Garmisch-Partenkirchen
  - "Nycomed Deutschland GmbH", Gebesee
  - "Nycomed Deutschland GmbH", Geisenhausen
  - "Nycomed Deutschland GmbH", Geislingen
  - "Nycomed Deutschland GmbH", Gelnhausen
  - "Nycomed Deutschland GmbH", Gelsenkirchen
  - "Nycomed Deutschland GmbH", Gemünden
  - "Nycomed Deutschland GmbH", Gensingen
  - "Nycomed Deutschland GmbH", Georgsmarienhütte
  - "Nycomed Deutschland GmbH", Gera
  - "Nycomed Deutschland GmbH", Gerbstedt
  - "Nycomed Deutschland GmbH", Geretsried
  - "Nycomed Deutschland GmbH", Gladbeck
  - "Nycomed Deutschland GmbH", Gladenbach
  - "Nycomed Deutschland GmbH", Glashütten
  - "Nycomed Deutschland GmbH", Gleichen
  - "Nycomed Deutschland GmbH", Glienicke
  - "Nycomed Deutschland GmbH", Goch
  - "Nycomed Deutschland GmbH", Goldberg
  - "Nycomed Deutschland GmbH", Göllingen
  - "Nycomed Deutschland GmbH", Görlitz
  - "Nycomed Deutschland GmbH", Gräfinau-Angstedt
  - "Nycomed Deutschland GmbH", Greiz
  - "Nycomed Deutschland GmbH", Greppin
  - "Nycomed Deutschland GmbH", Großaitingen
  - "Nycomed Deutschland GmbH", Großalmerode
  - "Nycomed Deutschland GmbH", Großburschla
  - "Nycomed Deutschland GmbH", Großefehn
  - "Nycomed Deutschland GmbH", Großhabersdorf
  - "Nycomed Deutschland GmbH", Großharthau-Bühlau
  - "Nycomed Deutschland GmbH", Großräschen
  - "Nycomed Deutschland GmbH", Großschirma
  - "Nycomed Deutschland GmbH", Grünbach
  - "Nycomed Deutschland GmbH", Grünheide
  - "Nycomed Deutschland GmbH", Gundelsheim
  - "Nycomed Deutschland GmbH", Güstrow
  - "Nycomed Deutschland GmbH", Hachenburg
  - "Nycomed Deutschland GmbH", Hadmersleben
  - "Nycomed Deutschland GmbH", Hagenow
  - "Nycomed Deutschland GmbH", Haigerloch
  - "Nycomed Deutschland GmbH", Halbe
  - "Nycomed Deutschland GmbH", Halberstadt
  - "Nycomed Deutschland GmbH", Haldensleben I
  - "Nycomed Deutschland GmbH", Halle
  - "Nycomed Deutschland GmbH", Hallstadt
  - "Nycomed Deutschland GmbH", Hamburg
  - "Nycomed Deutschland GmbH", Hamelin
  - "Nycomed Deutschland GmbH", Hamm
  - "Nycomed Deutschland GmbH", Hammelburg
  - "Nycomed Deutschland GmbH", Hanover
  - "Nycomed Deutschland GmbH", Harsewinkel
  - "Nycomed Deutschland GmbH", Hasbergen
  - "Nycomed Deutschland GmbH", Hauenstein
  - "Nycomed Deutschland GmbH", Hebertshausen
  - "Nycomed Deutschland GmbH", Heek
  - "Nycomed Deutschland GmbH", Heidelberg
  - "Nycomed Deutschland GmbH", Heilbad Heiligenstadt
  - "Nycomed Deutschland GmbH", Heilbronn
  - "Nycomed Deutschland GmbH", Helmstedt
  - "Nycomed Deutschland GmbH", Hemau
  - "Nycomed Deutschland GmbH", Hemmoor
  - "Nycomed Deutschland GmbH", Herborn
  - "Nycomed Deutschland GmbH", Herbrechtingen
  - "Nycomed Deutschland GmbH", Herbsleben
  - "Nycomed Deutschland GmbH", Herne
  - "Nycomed Deutschland GmbH", Herrnhut
  - "Nycomed Deutschland GmbH", Hesel
  - "Nycomed Deutschland GmbH", Hessisch Lichtenau
  - "Nycomed Deutschland GmbH", Hettstedt
  - "Nycomed Deutschland GmbH", Hilden
  - "Nycomed Deutschland GmbH", Hildesheim
  - "Nycomed Deutschland GmbH", Hirschaid
  - "Nycomed Deutschland GmbH", Hirschberg
  - "Nycomed Deutschland GmbH", Hirschfeld
  - "Nycomed Deutschland GmbH", Hofbieber
  - "Nycomed Deutschland GmbH", Hofheim
  - "Nycomed Deutschland GmbH", Hohenstein-Ernstthal
  - "Nycomed Deutschland GmbH", Höchheim
  - "Nycomed Deutschland GmbH", Husum
  - "Nycomed Deutschland GmbH", Hürth
  - "Nycomed Deutschland GmbH", Ibbenbueren
  - "Nycomed Deutschland GmbH", Ingolstadt
  - "Nycomed Deutschland GmbH", Jarmen
  - "Nycomed Deutschland GmbH", Jena
  - "Nycomed Deutschland GmbH", Jerichow
  - "Nycomed Deutschland GmbH", Jessen
  - "Nycomed Deutschland GmbH", Jettingen
  - "Nycomed Deutschland GmbH", Jever
  - "Nycomed Deutschland GmbH", Jockgrim
  - "Nycomed Deutschland GmbH", Jördenstorf
  - "Nycomed Deutschland GmbH", Jübek
  - "Nycomed Deutschland GmbH", Jüchen
  - "Nycomed Deutschland GmbH", Kaiserslautern
  - "Nycomed Deutschland GmbH", Kamen
  - "Nycomed Deutschland GmbH", Kamenz
  - "Nycomed Deutschland GmbH", Kandern
  - "Nycomed Deutschland GmbH", Kappeln
  - "Nycomed Deutschland GmbH", Karlsruhe
  - "Nycomed Deutschland GmbH", Kassel
  - "Nycomed Deutschland GmbH", Katzenelnbogen
  - "Nycomed Deutschland GmbH", Katzhütte
  - "Nycomed Deutschland GmbH", Kaufbeuren
  - "Nycomed Deutschland GmbH", Kelkheim
  - "Nycomed Deutschland GmbH", Kemnitz
  - "Nycomed Deutschland GmbH", Kempen
  - "Nycomed Deutschland GmbH", Kempenich
  - "Nycomed Deutschland GmbH", Kempten
  - "Nycomed Deutschland GmbH", Ketsch
  - "Nycomed Deutschland GmbH", Kevelaer
  - "Nycomed Deutschland GmbH", Kiefersfelden
  - "Nycomed Deutschland GmbH", Kiel
  - "Nycomed Deutschland GmbH", Kirchheimbolanden
  - "Nycomed Deutschland GmbH", Kleve
  - "Nycomed Deutschland GmbH", Klingenthal
  - "Nycomed Deutschland GmbH", Koblenz
  - "Nycomed Deutschland GmbH", Kolbermoor
  - "Nycomed Deutschland GmbH", Kolkwitz
  - "Nycomed Deutschland GmbH", Kornwestheim
  - "Nycomed Deutschland GmbH", Koßdorf
  - "Nycomed Deutschland GmbH", Kösching
  - "Nycomed Deutschland GmbH", Krefeld
  - "Nycomed Deutschland GmbH", Kreuztal
  - "Nycomed Deutschland GmbH", Kronach
  - "Nycomed Deutschland GmbH", Kronau
  - "Nycomed Deutschland GmbH", Kuchen
  - "Nycomed Deutschland GmbH", Kusterdingen
  - "Nycomed Deutschland GmbH", Künzing
  - "Nycomed Deutschland GmbH", Laage
  - "Nycomed Deutschland GmbH", Laatzen
  - "Nycomed Deutschland GmbH", Lahnau
  - "Nycomed Deutschland GmbH", Lalendorf
  - "Nycomed Deutschland GmbH", Lampertheim
  - "Nycomed Deutschland GmbH", Landau
  - "Nycomed Deutschland GmbH", Landshut
  - "Nycomed Deutschland GmbH", Langelsheim
  - "Nycomed Deutschland GmbH", Langenau
  - "Nycomed Deutschland GmbH", Langenbrettach
  - "Nycomed Deutschland GmbH", Langenhagen
  - "Nycomed Deutschland GmbH", Langenhessen
  - "Nycomed Deutschland GmbH", Langerwehe
  - "Nycomed Deutschland GmbH", Lauf
  - "Nycomed Deutschland GmbH", Lauingen
  - "Nycomed Deutschland GmbH", Lauterhofen
  - "Nycomed Deutschland GmbH", Lebach
  - "Nycomed Deutschland GmbH", Lehre
  - "Nycomed Deutschland GmbH", Leimen
  - "Nycomed Deutschland GmbH", Leipzig
  - "Nycomed Deutschland GmbH", Lemförde
  - "Nycomed Deutschland GmbH", Lengerich
  - "Nycomed Deutschland GmbH", Lensahn
  - "Nycomed Deutschland GmbH", Leverkusen
  - "Nycomed Deutschland GmbH", Lichtenfels
  - "Nycomed Deutschland GmbH", Limburgerhof
  - "Nycomed Deutschland GmbH", Lindow
  - "Nycomed Deutschland GmbH", Lommatzsch
  - "Nycomed Deutschland GmbH", Lorch
  - "Nycomed Deutschland GmbH", Löbejün
  - "Nycomed Deutschland GmbH", Löhne
  - "Nycomed Deutschland GmbH", Lubin
  - "Nycomed Deutschland GmbH", Ludwigsburg
  - "Nycomed Deutschland GmbH", Ludwigshafen
  - "Nycomed Deutschland GmbH", Lüdenscheid
  - "Nycomed Deutschland GmbH", Lügde
  - "Nycomed Deutschland GmbH", Lünen
  - "Nycomed Deutschland GmbH", Magdeburg
  - "Nycomed Deutschland GmbH", Mainz
  - "Nycomed Deutschland GmbH", Malchin
  - "Nycomed Deutschland GmbH", Mannheim
  - "Nycomed Deutschland GmbH", Marienheide
  - "Nycomed Deutschland GmbH", Markkleeberg
  - "Nycomed Deutschland GmbH", Marl
  - "Nycomed Deutschland GmbH", Marnitz
  - "Nycomed Deutschland GmbH", Matzlow-Garwitz
  - "Nycomed Deutschland GmbH", Mauer
  - "Nycomed Deutschland GmbH", Mayen
  - "Nycomed Deutschland GmbH", Meckenbeuren
  - "Nycomed Deutschland GmbH", Memmelsdorf
  - "Nycomed Deutschland GmbH", Menden
  - "Nycomed Deutschland GmbH", Mendig
  - "Nycomed Deutschland GmbH", Mengen
  - "Nycomed Deutschland GmbH", Mering
  - "Nycomed Deutschland GmbH", Merseburg
  - "Nycomed Deutschland GmbH", Mettmann
  - "Nycomed Deutschland GmbH", Metzingen
  - "Nycomed Deutschland GmbH", Mildstedt
  - "Nycomed Deutschland GmbH", Minden
  - "Nycomed Deutschland GmbH", Mittelherwigsdorf
  - "Nycomed Deutschland GmbH", Mittweida
  - "Nycomed Deutschland GmbH", Monheim
  - "Nycomed Deutschland GmbH", Monschau
  - "Nycomed Deutschland GmbH", Montabaur
  - "Nycomed Deutschland GmbH", Mönchengladbach
  - "Nycomed Deutschland GmbH", Murrhardt
  - "Nycomed Deutschland GmbH", Mühlhausen
  - "Nycomed Deutschland GmbH", Mülsen
  - "Nycomed Deutschland GmbH", München
  - "Nycomed Deutschland GmbH", Münchweiler
  - "Nycomed Deutschland GmbH", Münster
  - "Nycomed Deutschland GmbH", Nattheim
  - "Nycomed Deutschland GmbH", Nauen
  - "Nycomed Deutschland GmbH", Naumburg
  - "Nycomed Deutschland GmbH", Neckarbischofsheim
  - "Nycomed Deutschland GmbH", Neckargemünd
  - "Nycomed Deutschland GmbH", Neckarsulm
  - "Nycomed Deutschland GmbH", Neu Wulmstorf
  - "Nycomed Deutschland GmbH", Neu-Anspach
  - "Nycomed Deutschland GmbH", Neubrandenburg
  - "Nycomed Deutschland GmbH", Neufahrn
  - "Nycomed Deutschland GmbH", Neulußheim
  - "Nycomed Deutschland GmbH", Neumünster
  - "Nycomed Deutschland GmbH", Neunkirchen
  - "Nycomed Deutschland GmbH", Neuruppin
  - "Nycomed Deutschland GmbH", Neuss
  - "Nycomed Deutschland GmbH", Neustadt
  - "Nycomed Deutschland GmbH", Neustadt-Glewe
  - "Nycomed Deutschland GmbH", Neuwied
  - "Nycomed Deutschland GmbH", Niederlehme
  - "Nycomed Deutschland GmbH", Nienburg
  - "Nycomed Deutschland GmbH", Norderstedt
  - "Nycomed Deutschland GmbH", Nordhorn
  - "Nycomed Deutschland GmbH", Nordstemmen
  - "Nycomed Deutschland GmbH", Nossen
  - "Nycomed Deutschland GmbH", Nuremberg
  - "Nycomed Deutschland GmbH", Nünchritz
  - "Nycomed Deutschland GmbH", Oberdorla
  - "Nycomed Deutschland GmbH", Oberhausen
  - "Nycomed Deutschland GmbH", Oberkirch
  - "Nycomed Deutschland GmbH", Obertshausen
  - "Nycomed Deutschland GmbH", Oelsnitz
  - "Nycomed Deutschland GmbH", Oer-Erkenschwick
  - "Nycomed Deutschland GmbH", Oerel
  - "Nycomed Deutschland GmbH", Offenbach
  - "Nycomed Deutschland GmbH", Offstein
  - "Nycomed Deutschland GmbH", Oftersheim
  - "Nycomed Deutschland GmbH", Oldenburg
  - "Nycomed Deutschland GmbH", Oranienbaum
  - "Nycomed Deutschland GmbH", Oranienburg
  - "Nycomed Deutschland GmbH", Osloß
  - "Nycomed Deutschland GmbH", Osnabrück
  - "Nycomed Deutschland GmbH", Ostbevern
  - "Nycomed Deutschland GmbH", Osterburg
  - "Nycomed Deutschland GmbH", Ostritz
  - "Nycomed Deutschland GmbH", Ostseebad Kühlungsborn
  - "Nycomed Deutschland GmbH", Otterndorf
  - "Nycomed Deutschland GmbH", Overath
  - "Nycomed Deutschland GmbH", Paderborn
  - "Nycomed Deutschland GmbH", Panschwitz-Kuckau
  - "Nycomed Deutschland GmbH", Parchim
  - "Nycomed Deutschland GmbH", Passau
  - "Nycomed Deutschland GmbH", Peine
  - "Nycomed Deutschland GmbH", Petershagen
  - "Nycomed Deutschland GmbH", Pfullingen
  - "Nycomed Deutschland GmbH", Pfungstadt
  - "Nycomed Deutschland GmbH", Pinneberg
  - "Nycomed Deutschland GmbH", Plauen
  - "Nycomed Deutschland GmbH", Plön
  - "Nycomed Deutschland GmbH", Pockau
  - "Nycomed Deutschland GmbH", Porta Westfalica
  - "Nycomed Deutschland GmbH", Potsdam
  - "Nycomed Deutschland GmbH", Pößneck
  - "Nycomed Deutschland GmbH", Prüm
  - "Nycomed Deutschland GmbH", Pulsnitz
  - "Nycomed Deutschland GmbH", Radevormwald
  - "Nycomed Deutschland GmbH", Radis
  - "Nycomed Deutschland GmbH", Rastatt
  - "Nycomed Deutschland GmbH", Ratingen
  - "Nycomed Deutschland GmbH", Ravensburg
  - "Nycomed Deutschland GmbH", Redefin
  - "Nycomed Deutschland GmbH", Regensburg
  - "Nycomed Deutschland GmbH", Reichenbach
  - "Nycomed Deutschland GmbH", Reinbek
  - "Nycomed Deutschland GmbH", Rellingen
  - "Nycomed Deutschland GmbH", Remagen
  - "Nycomed Deutschland GmbH", Remscheid
  - "Nycomed Deutschland GmbH", Rendsburg
  - "Nycomed Deutschland GmbH", Reutlingen
  - "Nycomed Deutschland GmbH", Rheinberg
  - "Nycomed Deutschland GmbH", Rheine
  - "Nycomed Deutschland GmbH", Rodenbach
  - "Nycomed Deutschland GmbH", Rodewisch
  - "Nycomed Deutschland GmbH", Rohrbach
  - "Nycomed Deutschland GmbH", Rohrberg
  - "Nycomed Deutschland GmbH", Rosenfeld
  - "Nycomed Deutschland GmbH", Rostock
  - "Nycomed Deutschland GmbH", Rothenburg
  - "Nycomed Deutschland GmbH", Rottenburg
  - "Nycomed Deutschland GmbH", Rottleberode
  - "Nycomed Deutschland GmbH", Roßbach
  - "Nycomed Deutschland GmbH", Rösrath
  - "Nycomed Deutschland GmbH", Rudolstadt
  - "Nycomed Deutschland GmbH", Rülzheim
  - "Nycomed Deutschland GmbH", Rüsselsheim am Main
  - "Nycomed Deutschland GmbH", Saalburg-Ebersdorf
  - "Nycomed Deutschland GmbH", Saalfeld
  - "Nycomed Deutschland GmbH", Saint Blasien
  - "Nycomed Deutschland GmbH", Saint Georgen
  - "Nycomed Deutschland GmbH", Saint Ingbert
  - "Nycomed Deutschland GmbH", Salzkotten
  - "Nycomed Deutschland GmbH", Salzmünde
  - "Nycomed Deutschland GmbH", Sand
  - "Nycomed Deutschland GmbH", Sandesneben
  - "Nycomed Deutschland GmbH", Sangerhausen
  - "Nycomed Deutschland GmbH", Schellerten
  - "Nycomed Deutschland GmbH", Schenefeld
  - "Nycomed Deutschland GmbH", Schifferstadt
  - "Nycomed Deutschland GmbH", Schleswig
  - "Nycomed Deutschland GmbH", Schmelz
  - "Nycomed Deutschland GmbH", Schneeberg
  - "Nycomed Deutschland GmbH", Schollene
  - "Nycomed Deutschland GmbH", Schonungen
  - "Nycomed Deutschland GmbH", Schortens
  - "Nycomed Deutschland GmbH", Schönteichen
  - "Nycomed Deutschland GmbH", Schönwalde-Glien
  - "Nycomed Deutschland GmbH", Schriesheim
  - "Nycomed Deutschland GmbH", Schrobenhausen
  - "Nycomed Deutschland GmbH", Schwaig
  - "Nycomed Deutschland GmbH", Schwalbach
  - "Nycomed Deutschland GmbH", Schwalmstadt
  - "Nycomed Deutschland GmbH", Schwanewede
  - "Nycomed Deutschland GmbH", Schwarmstedt
  - "Nycomed Deutschland GmbH", Schwarzenbruck
  - "Nycomed Deutschland GmbH", Schwedt
  - "Nycomed Deutschland GmbH", Schweinitz
  - "Nycomed Deutschland GmbH", Schwerin
  - "Nycomed Deutschland GmbH", Schwetzingen
  - "Nycomed Deutschland GmbH", Seeheilbad Graal-Müritz
  - "Nycomed Deutschland GmbH", Selm
  - "Nycomed Deutschland GmbH", Seßlach
  - "Nycomed Deutschland GmbH", Sickte
  - "Nycomed Deutschland GmbH", Siegen
  - "Nycomed Deutschland GmbH", Silberstedt
  - "Nycomed Deutschland GmbH", Simmerath
  - "Nycomed Deutschland GmbH", Solingen
  - "Nycomed Deutschland GmbH", Sommerhausen
  - "Nycomed Deutschland GmbH", Sonneberg
  - "Nycomed Deutschland GmbH", Sömmerda
  - "Nycomed Deutschland GmbH", Spechbach
  - "Nycomed Deutschland GmbH", Speichersdorf
  - "Nycomed Deutschland GmbH", Speyer
  - "Nycomed Deutschland GmbH", Spiesen-Elversberg
  - "Nycomed Deutschland GmbH", Spremberg
  - "Nycomed Deutschland GmbH", Springe
  - "Nycomed Deutschland GmbH", Stadthagen
  - "Nycomed Deutschland GmbH", Stavenhagen
  - "Nycomed Deutschland GmbH", Steinfeld
  - "Nycomed Deutschland GmbH", Steinfurt
  - "Nycomed Deutschland GmbH", Stendal
  - "Nycomed Deutschland GmbH", Stockelsdorf
  - "Nycomed Deutschland GmbH", Stollberg
  - "Nycomed Deutschland GmbH", Stolpen
  - "Nycomed Deutschland GmbH", Strausberg
  - "Nycomed Deutschland GmbH", Stuhr
  - "Nycomed Deutschland GmbH", Stuttgart
  - "Nycomed Deutschland GmbH", Stützengrün
  - "Nycomed Deutschland GmbH", Suhl
  - "Nycomed Deutschland GmbH", Sulingen
  - "Nycomed Deutschland GmbH", Sulzbach
  - "Nycomed Deutschland GmbH", Tangermünde
  - "Nycomed Deutschland GmbH", Tarp
  - "Nycomed Deutschland GmbH", Taucha
  - "Nycomed Deutschland GmbH", Teterow
  - "Nycomed Deutschland GmbH", Thurnau
  - "Nycomed Deutschland GmbH", Timmendorfer Strand
  - "Nycomed Deutschland GmbH", Torgelow
  - "Nycomed Deutschland GmbH", Treffurt
  - "Nycomed Deutschland GmbH", Treis-Karden
  - "Nycomed Deutschland GmbH", Triebes
  - "Nycomed Deutschland GmbH", Tschernitz
  - "Nycomed Deutschland GmbH", Ueckermünde
  - "Nycomed Deutschland GmbH", Uelzen
  - "Nycomed Deutschland GmbH", Uffing
  - "Nycomed Deutschland GmbH", Uhlstädt-Kirchhasel
  - "Nycomed Deutschland GmbH", Ulm
  - "Nycomed Deutschland GmbH", Urbach
  - "Nycomed Deutschland GmbH", Vaihingen
  - "Nycomed Deutschland GmbH", Varel
  - "Nycomed Deutschland GmbH", Velbert
  - "Nycomed Deutschland GmbH", Viechtach
  - "Nycomed Deutschland GmbH", Viersen
  - "Nycomed Deutschland GmbH", Villingen-Schwenningen
  - "Nycomed Deutschland GmbH", Visselhövede
  - "Nycomed Deutschland GmbH", Vöhrenbach
  - "Nycomed Deutschland GmbH", Wagenfeld
  - "Nycomed Deutschland GmbH", Waiblingen
  - "Nycomed Deutschland GmbH", Waidhaus
  - "Nycomed Deutschland GmbH", Waldbröl
  - "Nycomed Deutschland GmbH", Wallerfing
  - "Nycomed Deutschland GmbH", Waltrop
  - "Nycomed Deutschland GmbH", Wannweil
  - "Nycomed Deutschland GmbH", Warstein
  - "Nycomed Deutschland GmbH", Wattenheim
  - "Nycomed Deutschland GmbH", Wegberg
  - "Nycomed Deutschland GmbH", Weibern
  - "Nycomed Deutschland GmbH", Weida
  - "Nycomed Deutschland GmbH", Weiden
  - "Nycomed Deutschland GmbH", Weilheim
  - "Nycomed Deutschland GmbH", Weinheim
  - "Nycomed Deutschland GmbH", Weinsberg
  - "Nycomed Deutschland GmbH", Weißenhorn
  - "Nycomed Deutschland GmbH", Weißwasser
  - "Nycomed Deutschland GmbH", Welden
  - "Nycomed Deutschland GmbH", Westerburg
  - "Nycomed Deutschland GmbH", Westerrönfeld
  - "Nycomed Deutschland GmbH", Wetter
  - "Nycomed Deutschland GmbH", Wetzlar
  - "Nycomed Deutschland GmbH", Wiehl
  - "Nycomed Deutschland GmbH", Wiesbaden
  - "Nycomed Deutschland GmbH", Willebadessen
  - "Nycomed Deutschland GmbH", Willich
  - "Nycomed Deutschland GmbH", Winkelhaid
  - "Nycomed Deutschland GmbH", Winsen
  - "Nycomed Deutschland GmbH", Wirges
  - "Nycomed Deutschland GmbH", Witten
  - "Nycomed Deutschland GmbH", Wittenberg
  - "Nycomed Deutschland GmbH", Wittlich
  - "Nycomed Deutschland GmbH", Wittstock
  - "Nycomed Deutschland GmbH", Woltersdorf
  - "Nycomed Deutschland GmbH", Worms
  - "Nycomed Deutschland GmbH", Wörnitz
  - "Nycomed Deutschland GmbH", Wörth
  - "Nycomed Deutschland GmbH", Wriedel
  - "Nycomed Deutschland GmbH", Wriezen
  - "Nycomed Deutschland GmbH", Wuppertal
  - "Nycomed Deutschland GmbH", Wurzen
  - "Nycomed Deutschland GmbH", Wustermark
  - "Nycomed Deutschland GmbH", Wustrau
  - "Nycomed Deutschland GmbH", Würzburg
  - "Nycomed Deutschland GmbH", Zarrentin
  - "Nycomed Deutschland GmbH", Zell
  - "Nycomed Deutschland GmbH", Zerbst
  - "Nycomed Deutschland GmbH", Zühlsdorf
  - "Nycomed Deutschland GmbH", Zweibrücken
  - "Nycomed Deutschland GmbH", Zwickau